CLINICAL TRIAL: NCT02015832
Title: Single-arm Trial Evaluating the Effectiveness of PCI of de Novo 3-vessel Disease Applying the SYNTAX Score II With Pressure Wire Functional Assessment and IVUS Guidance, Using an Everolimus-eluting Stent With Biodegradable Abluminal Coating
Brief Title: Trial Evaluating New Strategy in the Functional Assessment of 3-vessel Disease Using SYNTAXII Score in Patients With PCI
Status: Completed | Type: Observational
Sponsor: ECRI bv (Industry)
Collaborators: Boston Scientific Corporation (Industry); Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ECRI-002
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Heart Diseases; Cardiovascular Diseases; 3 Vessel Coronary Artery Disease
Keywords: SYNTAX II Score; Pressure wires; instantaneous wave-free ratio; fractional flow reserve; intravascular ultrasound; Drug eluting stents; Stents; Angioplasty; multi slice computed tomography
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Percutaneous Coronary Intervention: All patients (single arm study) will be receiving the SYNERGY™ Everolimus eluting stent (EES)
  Interventions: Device: Coronary stent; Radiation: Multi Slice Computed Tomography; Device: instantaneous wave-free ratio; Device: Fractional flow reserve; Device: Intravascular Ultrasound

INTERVENTIONS:
Device: Coronary stent
  Other Names: SYNERGY™ EES
Radiation: Multi Slice Computed Tomography — A coronary non-invasive Multi Slice Computed Tomography will be performed in patients
  Other Names: MSCT
Device: instantaneous wave-free ratio — Pressure-derived, adenosine-free index on physiological assessment of stenosis severity
  Other Names: iFR
Device: Fractional flow reserve — Pressure-derived index on physiological assessment of stenosis severity
  Other Names: FFR
Device: Intravascular Ultrasound — Allows the application of ultrasound technology to see from inside blood vessels out through the surrounding blood column, visualizing the inner wall of blood vessels
  Other Names: IVUS

SUMMARY:
Clinical study that aims to evaluate a new strategy using the SYNTAX II Score calculator in the functional assessment of patients with new coronary 3-vessel-disease who undergo percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
The purpose of the SYNTAX II Trial is to investigate the management of de-novo 3-vessel-disease in order to prospectively assess which patients would have at least comparable short and long term clinical outcomes between coronary artery bypass graft and percutaneous coronary intervention (PCI), using contemporary PCI practice. In SYNTAX II the effectiveness of a contemporary stent (designed with thinner struts, biocompatible and biodegradable polymer, and a limus based drug), the use of pressure wire assessment of lesions to allow for ischemia-driven revascularisation, intravascular ultrasound (IVUS) guidance to optimise drug eluting stent deployment, and the treatment of (chronic) total occlusion lesions with contemporary techniques, will be compared against PCI practice in the original SYNTAX trial. The proposed study would involve the SYNTAX Score II to prospectively recruit subjects on the grounds of patient safety

ELIGIBILITY:
Inclusion Criteria:

* At least 1 stenosis, angiographic, visually determined de novo lesions with more than 50 percent diameter stenosis in all 3 major epicardial territories. These are left descending coronary artery (LAD) and or side branch, proximal circumflex coronary artery (LCX) and or side branch, right descending coronary artery (RCA) and or side branch which are supplying viable myocardium without left main involvement. Patients with ostial LAD or ostial CX Medina 0,0,1 or Medina 0,1,0 may be enrolled
* Patients with hypoplastic RCA with absence of descending posterior and presence of a lesion in the LAD and CX territories may be included in the trial as a 3 vessel disease equivalent
* Vessel size should be at least 1.5 mm in diameter as visually assessed in diagnostic angiogram
* Patients with

  1. stable (Canadian Cardiovascular Society Class 1, 2, 3 or 4) angina pectoris
  2. or unstable (Braunwald class) angina pectoris and ischemia
  3. or patients with atypical chest pain or those who are asymptomatic provided they have myocardial ischemia, for example treadmill exercise test, radionuclide scintigraphy, stress echocardiography
* All anatomical SYNTAX Scores are eligible for initial screening with the SYNTAX Score II
* Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site
* Signed Heart Team Decision Form between local cardiologist and surgeon that the selected case meets all of the inclusion and exclusion criteria

Exclusion Criteria:

* Under the age of 21 years
* Known pregnancy at time of enrolment. Female of childbearing potential, and last menstruation within the last 12 months, who are not taking adequate contraceptives. Female who is breastfeeding at time of enrolment
* Prior PCI or CABG
* Ongoing acute myocardial infarction and enzymes (CKMB) more than 2x upper limit of normal
* Concomitant cardiac valve disease requiring surgical therapy, reconstruction or replacement
* Single or two-vessel disease at time of Heart Team consensus
* Participation or planned participation in another cardiovascular clinical study before one year follow up is completed
* Mental condition, psychiatric or organ cerebral disease, rendering the subject unable to understand the nature, scope, and possible consequences of the study or mental retardation or language barrier such that the patient is unable to give informed consent and potential for non-compliance towards the requirement in the study protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with de novo 3 vessel disease
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Spitzer, MD, Study Director — European Cardiovascular Research Institute; Javier Escaned, MD, Principal Investigator — Hospital San Carlos Madrid, Spain; Adrian Banning, MD, Principal Investigator — John Radcliffe Hospital, Oxford, United Kingdom
Locations (22):
- Netherlands (2):
  - Research Center NL007, Amsterdam, North Holland
  - Research Center NL001, Rotterdam, South Holland
- Poland (4):
  - Research Center PL008, Bielsko-Biala
  - Research Center PL012, Katowice
  - Research Center PL010, Krakow
  - Research Center PL004, Poznan
- Spain (7):
  - Research Center ES009, Santander, Cantabria
  - Research Center ES001, Barcelona, Catalonia
  - Research Center ES004, Vigo, Galicia
  - Research Center ES007, Madrid, Madrid
  - Research Center ES012, Madrid, Madrid
  - Research Center ES015, Madrid, Madrid
  - Research Center ES016, Salamanca
- United Kingdom (9):
  - Research Center GB014, Belfast, County Antrim
  - Research Center GB019, Oxford, Oxfordshire
  - Research Center GB005, Brighton
  - Research Center GB020, Cambridge
  - Research Center GB015, Edinburgh
  - Research Center GB001, Liverpool
  - Research Center GB017, London
  - Research Center GB006, Manchester
  - Research Center GB013, Newcastle upon Tyne

REFERENCES:
- [Derived] Wang R, Kawashima H, Hara H, Gao C, Ono M, Takahashi K, Tu S, Soliman O, Garg S, van Geuns RJ, Tao L, Wijns W, Onuma Y, Serruys PW. Comparison of Clinically Adjudicated Versus Flow-Based Adjudication of Revascularization Events in Randomized Controlled Trials. Circ Cardiovasc Qual Outcomes. 2021 Nov;14(11):e008055. doi: 10.1161/CIRCOUTCOMES.121.008055. Epub 2021 Oct 20. PMID 34666500
- [Derived] Collet C, Miyazaki Y, Ryan N, Asano T, Tenekecioglu E, Sonck J, Andreini D, Sabate M, Brugaletta S, Stables RH, Bartorelli A, de Winter RJ, Katagiri Y, Chichareon P, De Maria GL, Suwannasom P, Cavalcante R, Jonker H, Morel MA, Cosyns B, Kappetein AP, Taggart DT, Farooq V, Escaned J, Banning A, Onuma Y, Serruys PW. Fractional Flow Reserve Derived From Computed Tomographic Angiography in Patients With Multivessel CAD. J Am Coll Cardiol. 2018 Jun 19;71(24):2756-2769. doi: 10.1016/j.jacc.2018.02.053. Epub 2018 May 22. PMID 29802016
- [Derived] Escaned J, Collet C, Ryan N, De Maria GL, Walsh S, Sabate M, Davies J, Lesiak M, Moreno R, Cruz-Gonzalez I, Hoole SP, Ej West N, Piek JJ, Zaman A, Fath-Ordoubadi F, Stables RH, Appleby C, van Mieghem N, van Geuns RJ, Uren N, Zueco J, Buszman P, Iniguez A, Goicolea J, Hildick-Smith D, Ochala A, Dudek D, Hanratty C, Cavalcante R, Kappetein AP, Taggart DP, van Es GA, Morel MA, de Vries T, Onuma Y, Farooq V, Serruys PW, Banning AP. Clinical outcomes of state-of-the-art percutaneous coronary revascularization in patients with de novo three vessel disease: 1-year results of the SYNTAX II study. Eur Heart J. 2017 Nov 7;38(42):3124-3134. doi: 10.1093/eurheartj/ehx512. PMID 29020367
- [Derived] Farooq V, Serruys PW. Bypass Grafting Versus Percutaneous Intervention-Which Is Better in Multivessel Coronary Disease: Lessons From SYNTAX and Beyond. Prog Cardiovasc Dis. 2015 Nov-Dec;58(3):316-34. doi: 10.1016/j.pcad.2015.10.002. Epub 2015 Oct 31. PMID 26529569

RESULTS

PARTICIPANT FLOW:
Groups:
- Percutaneous Coronary Intervention: All-Comers, angiographic, de-novo 3-vessel disease without left main involvement (visual % diameter stenosis #50%).
Period: Overall Study
Arm/Group | Percutaneous Coronary Intervention
Started | 454
Completed | 443
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 423
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 36
  Poland | 38
  United Kingdom | 230
  Spain | 150

OUTCOME MEASURES:

1. Primary Outcome: Umber of Participants With Major Adverse Cardiac and Cerebrovascular Events (MACCE)
Description: MACCE is defined as: all-cause death; cerebrovascular event (stroke); documented myocardial infarction or all-cause revascularization
Time Frame: 1 year
Population: All patients enrolled in the SYNTAX II single-arm study were compared with a historical cohort selected from the SYNTAX I PCI arm (NCT00114972). Patients had three-vessel disease at presentation and qualified to enter the study based on equipoise to undergo either PCI or CABG according to the SYNTAX score II calculator (www.syntaxscore.org).
Measure: Count of Participants; unit: Participants
Groups:
- SYNTAX II PCI Strategy Arm: Use of the SYNTAX II PCI strategy in patients with de novo three vessel disease. SYNTAX II PCI strategy included use of new generation DES, coronary physiology, and coronary imaging for stent implantation.
- Pre-defined SYNTAX I PCI Cohort: The historical comparator consisted on subjects enrolled in the SYNTAX I trial, treated with PCI, who would fulfill the SYNTAX II score criteria used in SYNTAX II (i.e. similar risk of undergoing PCI or CABG based on predicted mortality at 4 years).
Arm/Group | SYNTAX II PCI Strategy Arm | Pre-defined SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 47 | 54

2. Secondary Outcome: Number of Participants With All-cause Death, Stroke, or Myocardial Infarction
Description: Safety endpoint
Time Frame: 1 Year
Population: SYNTAX II PCI cohort vs. SYNTAX I PCI selected cohort.
Measure: Count of Participants; unit: Participants
Groups:
- SYNTAX II PCI Cohort: Patient with de-novo three vessel disease undergoing PCI according to the SYNTAX II strategy, including coronary physiology, imaging, and new generation drug-eluting stents.
- SYNTAX I PCI Cohort: Patient with de-novo three vessel disease undergoing PCI according in the SYNTAX I trial, who would qualify as comparators for SYNTAX II based on equipoise between CABG and PCI using the SYNTAX score II calculator (www.syntaxscore.org).
Arm/Group | SYNTAX II PCI Cohort | SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 17 | 20

3. Secondary Outcome: Number of Participants With All-cause Death
Description: All-cause death
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Groups:
- SYNTAX II PCI Cohort: Patients with de-novo three vessel disease undergoing PCI according to the SYNTAX II strategy, including coronary physiology, imaging, and new generation drug-eluting stents.
- SYNTAX I PCI Cohort: Patients with de-novo three vessel disease undergoing PCI according in the SYNTAX I trial, who would qualify as comparators for SYNTAX II based on equipoise between CABG and PCI using the SYNTAX score II calculator (www.syntaxscore.org).
Arm/Group | SYNTAX II PCI Cohort | SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 9 | 9

4. Secondary Outcome: Number of Participants With Stroke
Description: Stroke
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | SYNTAX II PCI Cohort | SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 2 | 2

5. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: Any myocardial infarction
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SYNTAX II PCI Cohort | SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 6 | 15

6. Secondary Outcome: Number of Participants With Revascularization
Description: Any coronary revascularization
Time Frame: 1 Years
Measure: Count of Participants; unit: Participants
Arm/Group | SYNTAX II PCI Cohort | SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 36 | 42

7. Secondary Outcome: Number of Participants With Definite Stent Thrombosis
Description: Stent Thrombosis - according to ARC definitions. Definite ST can be confirmed with 1) angiography (the presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent and presence of at least 1 of the following criteria within a 48-hour time window: Acute onset of ischemic symptoms at rest; New ischemic ECG changes that suggest acute ischemia; Typical rise and fall in cardiac biomarkers (refer to definition of spontaneous MI); Non-occlusive thrombus or Occlusive thrombus; or 2) Pathological confirmation (evidence of recent thrombus within the stent determined at autopsy or via examination of tissue retrieved following thrombectomy).
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | SYNTAX II PCI Cohort | SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 3 | 8

8. Secondary Outcome: Number of Participants With Probable Stent Thrombosis
Description: Stent Thrombosis - according to ARC definitions. Clinical definition of probable stent thrombosis is considered to have occurred after intracoronary stenting in the following cases: 1) Any unexplained death within the first 30 days; 2) Irrespective of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SYNTAX II PCI Cohort | SYNTAX I PCI Cohort
Number analyzed (Participants) | 454 | 315
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Percutaneous Coronary Intervention
All-Cause Mortality (participants affected / at risk) | 36/454
Serious Adverse Events (participants affected / at risk) | 125/454
Other Adverse Events (participants affected / at risk) | 0/454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Coronary Intervention (N=454)
Myocardial Infarction (Cardiac disorders) | 12 (125)
All-cause Revascularization (Cardiac disorders) | 60 (125)
Stroke (Cardiac disorders) | 10 (125)
Stent Thrombosis (Cardiac disorders) | 7 (125)
Death (General disorders) | 36 (125)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT02015832/Prot_SAP_000.pdf